CLINICAL TRIAL: NCT01331499
Title: A Post-Market, Prospective, Multicenter, Randomized Trial Comparing the Use of Standard of Care Blood Sparing Techniques With and Without the Aquamantys System to Facilitate Hemostasis in Subjects Undergoing Multi-level Spinal Fusions
Brief Title: Salient Aquamantys Spine Trial
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study terminated due to Medtronic acquisition
Sponsor: Salient Surgical Technologies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SAL-SP-10-001
Record Dates: First submitted 2011-04-06; First posted 2011-04-08 (Estimated); Last update posted 2012-06-07 (Estimated); Status verified 2012-06

CONDITIONS: Blood Loss
Keywords: Blood loss; transfusions; instrumented spinal fusion
MeSH Terms: conditions — Hemorrhage | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bipolar Sealer (Experimental): Standard of care blood sparing techniques with bipolar sealer
  Interventions: Device: Bipolar Sealer (Aquamantys)
- Control (Active Comparator): Standard of care blood sparing techniques without the use of bipolar sealer
  Interventions: Procedure: Standard of Care

INTERVENTIONS:
Device: Bipolar Sealer (Aquamantys) — Standard of care blood sparing techniques along with the use of bipolar sealer
  Other Names: Aquamantys
  Arms: Bipolar Sealer
Procedure: Standard of Care — Standard of care blood sparing techniques without the useof bipolar sealer
  Arms: Control

SUMMARY:
The purpose of this study is to compare standard of care hemostasis techniques with and without the use of Aquamantys in reducing peri-operative blood loss.

DETAILED DESCRIPTION:
The primary objective of the study is to assess the effectiveness of Aquamantys in reducing peri-operative blood loss compared with standard electrocautery

Secondary objectives include :

* Rate and volume of transfusions
* Evaluating the reduction in hemoglobin and hematocrit values post- operatively
* LOS costs, and operative time
* Gathering operator feedback on qualitative criteria, including ease of use and surgical visualization between the two treatment groups

ELIGIBILITY:
Inclusion Criteria:

1. Be candidate for three level (or greater) fusion surgery from T1 to S1 utilizing a direct posterior approach
2. Male or female 18 to 70 years of age (inclusive)
3. Must sign the IRB approved Informed Consent Form

Exclusion Criteria:

1. Undergoing spinal fusion for < 3 lumbar levels, or using an approach other than direct posterior
2. Undergoing an interbody fusion
3. Planned use of hypotensive anaesthesia
4. Pregnant or lactating
5. Morbid obesity, defined as Body Mass Index (BMI) greater than 40
6. Previously diagnosed coagulopathy or bleeding diasthesis
7. Currently, or within the previous 7 days prior to surgery, taking any medications that would produce bleeding diathesis including, but not limited to NSAIDs, aspirin, clopidogrel (Plavix), ticlopidine, or valproic acid
8. History of significant cardiac disorders that would necessitate special fluid management protocols
9. Serious trauma other than that confined to the spine
10. History of acute myocardial infarction and/or acute angina within the past year prior to enrollment
11. PT/INR >1.3 in the 14 days prior to surgery
12. PTT > 40 in the 14 days prior to surgery
13. Platelet count <100K in the 14 days prior to surgery
14. Based on clinical history, physical exam and subject presentation, subject has or is suspected to have a history of alcohol and/or drug abuse that would preclude subject from providing adequate consent and/or complying with study requirements
15. Prisoner or transient
16. Enrolled in another drug or device investigational study (currently or within past 30 days)
17. Unable or unwilling to sign the Informed Consent Form or comply with protocol specified procedures

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-04; Primary Completion 2012-12 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Actual Peri-operative Blood Loss | Up to 72 hours post-operatively
  Actual blood loss (ABL) will be calculated using a study specified formula using laboratory data from up to 72 hours post-surgery. ABL will be compared between treatment groups

SECONDARY OUTCOMES:
Frequency and volume of transfusions | Up to 72 hours post-operatively
  The frequency and volume of transfusions will be measured between treatment groups
Reduction in hemoglobin and hematocrit values post-operatively | Upto 72 hours post-operatively
  The reduction in hemoglobin and hematocrit values will be evaluated between the two treatment groups
Length of stay costs and operativ time | Up to 21 days post-operatively
  Total length of staycosts and operative time will be compared between treatment groups.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Fischgrund, M.D., Principal Investigator — Corewell Health East
Locations (3):
- United States (3):
  - George Washington University Medical Center, Washington D.C., District of Columbia
  - Rush University Medical Center, Chicago, Illinois
  - William Beaumont Hospital, Royal Oak, Michigan